CLINICAL TRIAL: NCT00104286
Title: An Open-Label, Single-Arm, Phase I Study of Troxatyl™ (Troxacitabine) Administered by Continuous Infusion in Subjects With an Advanced Solid Malignancy
Brief Title: Study of Troxatyl™ Administered by Continuous Infusion to Subjects With Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SGX Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD758-109
Record Dates: First submitted 2005-02-24; First posted 2005-02-25 (Estimated); Last update posted 2006-11-03 (Estimated); Status verified 2006-11

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — troxacitabine

INTERVENTIONS:
Drug: Troxatyl™ (Cytotoxic Chemotherapeutic)

SUMMARY:
This is a phase I, single-arm, open-label, single-center study to establish the recommended infusion schedule for Troxatyl™ administered as a continuous infusion for 2-5 days to subjects with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced solid malignancy refractory to prior therapy and unlikely to benefit from known therapies (e.g., chemotherapy, radiation therapy, and surgery).
* Diagnosis confirmed histologically or cytologically.
* Subjects may have received prior cancer therapy (including surgery, radiotherapy, chemotherapy, and hormonal therapy), but must have completed all therapies at least 30 days prior to study drug administration (42 days for nitrosourea or mitomycin).
* Subjects must have recovered from the toxic effects associated with prior treatment.
* Subjects must have an Eastern Cooperative Oncology Group performance status of ≤ 2 and an estimated life expectancy of at least 12 weeks.
* Subjects must have adequate organ and immune function as indicated by standard laboratory tests.
* The subject must understand, be able, willing, and likely to fully comply with study procedures, including scheduled follow-up, and restrictions.
* The subject must give written, personally signed and dated, informed consent to participate in the study before implementing any study related procedures.

Exclusion Criteria:

* Previously documented brain metastases.
* Active and uncontrolled infection.
* Subjects with uncontrolled medical problems, unrelated to the malignancy, or of sufficient severity that in the opinion of the investigator, impair their ability to give informed consent or unacceptably reduce the safety of the proposed treatment.
* Neurological or psychiatric disorders that would interfere with consent or study follow-up.
* Prior treatment with more than 6 courses of alkylating agent-containing chemotherapy (except low-dose cisplatin) or more than 4 courses of carboplatin, radiation therapy to > 25% of hematopoietic reserves or two or more courses of mitomycin C or nitrosourea.
* Known or suspected intolerance or hypersensitivity to the study materials [or closely related compounds] or any of their stated ingredients.
* History of alcohol or other substance abuse within the last year.
* Use of another investigational agent or participation in a clinical trial within 30 days prior to enrollment.
* Female subjects who are pregnant or lactating, including females with a positive pregnancy test at screening must be excluded.
* Subjects that have previously been enrolled into this study and subsequently withdrawn must also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-01; Study Completion 2005-11

PRIMARY OUTCOMES:
To determine the recommended infusion schedule for the investigational new drug administered as a continuous infusion, and to define the safety tolerance and dose limiting toxicities.

SECONDARY OUTCOMES:
Pharmacokinetic/pharmacodynamic profile, preliminary evidence of the anti-tumor activity.

CONTACTS AND LOCATIONS:
Locations (1):
- The Sydney Kimmel Comprehensive Cancer Center at John Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Background] Giles FJ. Troxacitabine-based therapy of refractory leukemia. Expert Rev Anticancer Ther. 2002 Jun;2(3):261-6. doi: 10.1586/14737140.2.3.261. PMID 12113049